CLINICAL TRIAL: NCT03525600
Title: A Phase 3, Multi-Center, Randomized, Double-Masked, Sham-Controlled Study to Compare the Efficacy and Safety of Intravitreal Pegcetacoplan Therapy With Sham Injections in Patients With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: Study to Compare the Efficacy and Safety of Intravitreal APL-2 Therapy With Sham Injections in Patients With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APL2-303
Record Dates: First submitted 2018-04-20; First posted 2018-05-15 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- APL-2 15mg 0.1 mL monthly for 24 months (Experimental): A single dose of 15 mg APL-2/0.1 mL will be administered via intravitreal injection in this study. Subjects will receive an injection every month
  Interventions: Drug: APL-2
- APL-2 15mg 0.1 mL EOM for 24 months (Experimental): A single dose of 15 mg APL-2/0.1 mL will be administered via intravitreal injection in this study. Subjects will receive an injection every other month
  Interventions: Drug: APL-2
- Sham Procedure Monthly for 24 months (Experimental): Sham Procedure for 24 months
  Interventions: Other: Sham Procedure
- Sham Procedure Every Other Month for 24 months (Experimental): Sham Procedure every other month for 24 months
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Drug: APL-2 — Complement (C3) Inhibitor
  Arms: APL-2 15mg 0.1 mL monthly for 24 months
Drug: APL-2 — Complement (C3) Inhibitor
  Arms: APL-2 15mg 0.1 mL EOM for 24 months
Other: Sham Procedure — Subjects will receive a Sham procedure every month
  Arms: Sham Procedure Monthly for 24 months
Other: Sham Procedure — Subjects will receive a Sham procedure every other month
  Arms: Sham Procedure Every Other Month for 24 months

SUMMARY:
This is a 24-month, Phase III, multicenter, randomized, double-masked, sham-injection controlled study to assess the efficacy and safety of multiple IVT injections of APL-2 in subjects with GA secondary to AMD.

ELIGIBILITY:
Inclusion Criteria:

The study eye must meet all inclusion criteria. If both eyes meet the inclusion criteria, the eye with the worst visual acuity at the screening visit will be designated as the study eye. If both eyes have the same visual acuity, the right eye will be selected as the study eye.

Ocular- specific inclusion criteria apply to the study eye only, unless otherwise specified.

* Age ≥ 60 years.
* Normal Luminance best corrected visual acuity of 24 letters or better using Early Treatment Diabetic Retinopathy Study (ETDRS) charts (approximately 20/320 Snellen equivalent).
* Clinical diagnosis of GA of the macula secondary to AMD as determined by the Investigator and confirmed by the Reading Center.
* The GA lesion must meet the following criteria as determined by the central reading center's assessment of Fundus Autofluorescence (FAF) imaging at screening:

  * Total GA area must be ≥ 2.5 and ≤ 17.5 mm2 (1 and 7 disk areas [DA] respectively)
  * If GA is multifocal, at least one focal lesion must be ≥ 1.25 mm2 (0.5 DA), with the overall aggregate area of GA as specified above in 4a.
  * The entire GA lesion must be completely visualized on the macula centered image and must be able to be imaged in its entirety and not contiguous with any areas of peripapillary atrophy.
  * Presence of any pattern of hyperautofluorescence in the junctional zone of GA. Absence of hyperautofluorescence (i.e. pattern = none) is exclusionary.
* Adequate clarity of ocular media, adequate pupillary dilation, and fixation to permit the collection of good quality images as determined by the Investigator.
* Female subjects must be:

  * Women of non-child-bearing potential (WONCBP), or
  * Women of child-bearing potential (WOCBP) with a negative serum pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study and refrain from breastfeeding for the duration of the study.
* Males with female partners of child-bearing potential must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study.
* Willing and able to give informed consent and to comply with the study procedures and assessments.

Exclusion Criteria:

Ocular specific exclusion criteria apply to the study eye only, unless otherwise specified.

* GA secondary to a condition other than AMD such as Stargardt disease, cone rod dystrophy or toxic maculopathies like plaquenil maculopathy in either eye.
* Spherical equivalent of the refractive error demonstrating > 6 diopters of myopia or an axial length >26 mm.
* Any history or active choroidal neovascularization (CNV), associated with AMD or any other cause, including any evidence of retinal pigment epithelium rips or evidence of neovascularization anywhere based on SD-OCT imaging and/or fluorescein angiography as assessed by the Reading Center.
* Presence of an active ocular disease that in the opinion of the Investigator compromises or confounds visual function, including but not limited to, uveitis, other macular diseases (e.g. clinically significant epiretinal membrane (ERM), full thickness macular hole or uncontrolled glaucoma/ocular hypertension. Benign conditions in the opinion of the investigator such as peripheral retina dystrophy are not exclusionary).
* Intraocular surgery (including lens replacement surgery) within 3 months prior to randomization.
* History of laser therapy in the macular region.
* Aphakia or absence of the posterior capsule. Note: YAG laser posterior capsulotomy for posterior capsule opacification done at least 60 days prior to screening is not exclusionary.
* Any ocular condition other than GA secondary to AMD that may require surgery or medical intervention during the study period or, in the opinion of the Investigator, could compromise visual function during the study period.
* Any contraindication to IVT injection including current ocular or periocular infection.
* History of prior intravitreal injection.
* Prior participation in another interventional clinical study for intravitreal therapies in either eye (including subjects receiving sham).
* Prior participation in another interventional clinical study for geographic atrophy in either eye including investigational oral medication and placebo.
* Participation in any systemic experimental treatment or any other systemic investigational new drug within 6 weeks or 5 half-lives of the active ingredient (whichever is longer) prior to the start of study treatment. Note: clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary.
* Medical or psychiatric conditions that, in the opinion of the investigator, make consistent follow-up over the 24-month treatment period unlikely, or would make the subject an unsafe study candidate.
* Any screening laboratory value (hematology, serum chemistry or urinalysis) that in the opinion of the Investigator is clinically significant and not suitable for study participation.
* Known hypersensitivity to fluorescein sodium for injection or hypersensitivity to APL-2 or any of the excipients in APL-2 solution.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (141):
- United States (73):
  - Retinal Research Institute, Phoenix, Arizona
  - Associated Retina Consultants, Ltd, Phoenix, Arizona
  - Retina Institute of California dba Acuity Eye Grp, Arcadia, California
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - The Gavin Herbert Eye Institute/UC Irvine, Irvine, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Institute of California Medical Group, Palm Desert, California
  - Byers Eye Institute at Standford, Stanford School of Medicine, Palo Alto, California
  - Retina Consultants San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Danbury Eye Physicians & Surgeons, P.C. - Danbury, Danbury, Connecticut
  - New England Retina Associates, Hamden, Connecticut
  - Retina Group of New England,PC, Waterford, Connecticut
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Pinnacle Research Institute, Fort Lauderdale, Florida
  - Retina Health Center, Fort Myers, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Retina Associates of Florida, Tampa, Florida
  - University of South Florida (USF) Eye Institute, Tampa, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Georgia Retina, Marietta, Georgia
  - Midwest Eye Institute, Indianapolis, Indiana
  - Sabates Eye Center, Leawood, Kansas
  - Elman Retina Group, PA, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, PC, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Retina Specialists, Towson, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants, PC, Springfield, Massachusetts
  - Associated Retinal Consultants, P.C, Grand Rapids, Michigan
  - Retina Specialists of Michigan / Foundation for Vision, Grand Rapids, Michigan
  - Retina Consultants of Michigan, Southfield, Michigan
  - Associated Retinal Consultants PC, Traverse City, Michigan
  - Sierra Eye Associates, Reno, Nevada
  - Retina Associates of New Jersey (NJ Retina), Teaneck, New Jersey
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Vitreous Retina Macula Consultants of NY, New York, New York
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates, PS, Charlotte, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - Retina Associates of Cleveland, Inc., Cleveland, Ohio
  - Retina Associates of Cleveland, Inc, Cleveland, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cole Eye Institute, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Retina Associates of Cleveland, Inc., Youngstown, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Eye Health Northwest, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Southwest Retina Specialists, Amarillo, Texas
  - Retina Consultants of Austin (Retina Research Center), Austin, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Retina Associates of Utah, PC, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - The Retina Group of Washington, Fairfax, Virginia
  - Virginia Retina Center, Warrenton, Virginia
  - Vitreoretinal Associates of Washington, Bellevue, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (10):
  - Fundacion Zambrano, Buenos Aires, Buenos Aires F.D.
  - Microcirugia Ocular, El Rosario, Corrientes Province
  - Grupo Laser Vision, Rosario, Santa Fe Province
  - Organizacion Medica de investigacion, Buenos Aires
  - Centro Oftalmologico Dr Charles, Buenos Aires
  - Diagnostico Ocular, Buenos Aires
  - Centro Privado de Ojos Romagosa SA, Córdoba
  - Instituto Oftalmologico de Cordoba, Córdoba
  - Oftar Mendoza SRL, Mendoza
  - Oftalmologos Especialistas, Rosario
- Australia (3):
  - Sydney Retina, Sydney, New South Wales
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Retina and Eye Consultants, Hurstville
- Brazil (6):
  - Clinica Ocular Oftalmologia LTDA, Vitória, Espírito Santo
  - Clinica Oftalmologica Sao Lucas, Osasco, São Paulo
  - IPEPO - Instituto Da Visao, São Paulo, Vila Clementino
  - Instituto da Visão - Hospital de Olhos Ltda, Belo Horizonte
  - Hospital De Clinicas De Porto Alegre, Porto Alegre
  - UNIFESP - Federal University, São Paulo
- Canada (4):
  - Ivey Eye Institute, London, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - DRY AMD Clinic - St. Michael's Hospital, Toronto, Ontario
  - Retina Centre of Ottawa, Ottawa
- Czechia (4):
  - University Hospital Kralovske Vinochrady, Brno-Vinohrady
  - Fakultní nemocnice Ostrava, Ostrava-Poruba
  - OFTEX Eye Clinic, Pardubice
  - AXON Clinical, S.R.O., Prague
- France (7):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hopital de la Croix-Rousse, Lyon
  - Centre Monticelli Paradis, Marseille
  - CHU de Nantes - Hotel Dieu, Nantes
  - Centre Ophtalmologique de l´Odéon, Paris
  - Centre Ophthalmologique Saint-Exupery, Saint-Cyr-sur-Loire
  - Maison Rouge Ophthalmologic Center, Strasbourg
- Germany (6):
  - Universitäts-Augenklinik Bonn, Bonn
  - University Hospital Cologne, Cologne
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Klinikum rechts der Isar, München
  - Universitätsklinikum Regensburg, Regensburg
  - University Hospital Würzburg, Würzburg
- Israel (6):
  - Shamir Medical Center, Be’er Ya‘aqov
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Luigi Sacco Hospital, Milan
- New Zealand (2):
  - Retina Specialist, Auckland
  - Hamilton Eye Clinic, Hamilton
- Poland (4):
  - Oftalmika Eye Hospital, Bydgoszcz
  - Jasne Blonia Eye Clinic, Lodz
  - Centrum Diagnostyki i Mikrochirurgii Oka - LENS, Olsztyn
  - Centrum Medyczne UNO-MED, Tarnów
- Emanuelli Research and Development Center, Arecibo, Puerto Rico
- Spain (3):
  - Centro Médico Teknon, Barcelona
  - Instituto Oftalmologico Gómez-Ulla, Santiago de Compostela
  - Hospital Universitario Rio Hortega, Valladolid
- United Kingdom (10):
  - Moorfields Eye Hospital NHS Foundation Trust, London, England
  - Eye Clinic, Acre Mill Outpatients, Huddersfield Royal Infirmary, Huddersfield, West Yorkshire
  - Bristol Eye Hospital, Bristol
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - London North West University Hospital Trust, London
  - King's College Hospital NHS Trust, London
  - Oxford Eye Hospital, Oxford
  - Salisbury NHS Foundation Trust, Salisbury
  - Sunderland Eye Infirmary, Sunderland

REFERENCES:
- [Derived] Sadda S, Hatcher KA, Shah BK, Kondapalli SS, Li C, Baumal CR. Outer Retinal Tubulation and Geographic Atrophy: A Natural History Analysis of Sham Observed Eyes from the OAKS and DERBY Trials. Ophthalmol Ther. 2025 Jul;14(7):1611-1619. doi: 10.1007/s40123-025-01156-5. Epub 2025 May 19. PMID 40388106
- [Derived] Wykoff CC, Holz FG, Chiang A, Boyer D, Dhoot DS, Loewenstein A, Mones J, Heier J, Abbey AM, Singerman LJ, Vajzovic L, Lin J, Li C, Vilupuru A, Baumal CR; OAKS, DERBY, and GALE Investigators. Pegcetacoplan Treatment for Geographic Atrophy in Age-Related Macular Degeneration Over 36 Months: Data From OAKS, DERBY, and GALE. Am J Ophthalmol. 2025 Aug;276:350-364. doi: 10.1016/j.ajo.2025.04.016. Epub 2025 Apr 23. PMID 40280279
- [Derived] Fu DJ, Bagga P, Naik G, Glinton S, Faes L, Liefers B, Lima R, Wignall G, Keane PA, Ioannidou E, Ribeiro Reis AP, McKeown A, Scheibler L, Patel PJ, Moghul I, Pontikos N, Balaskas K. Pegcetacoplan Treatment and Consensus Features of Geographic Atrophy Over 24 Months. JAMA Ophthalmol. 2024 Jun 1;142(6):548-558. doi: 10.1001/jamaophthalmol.2024.1269. PMID 38722644
- [Derived] Heier JS, Lad EM, Holz FG, Rosenfeld PJ, Guymer RH, Boyer D, Grossi F, Baumal CR, Korobelnik JF, Slakter JS, Waheed NK, Metlapally R, Pearce I, Steinle N, Francone AA, Hu A, Lally DR, Deschatelets P, Francois C, Bliss C, Staurenghi G, Mones J, Singh RP, Ribeiro R, Wykoff CC; OAKS and DERBY study investigators. Pegcetacoplan for the treatment of geographic atrophy secondary to age-related macular degeneration (OAKS and DERBY): two multicentre, randomised, double-masked, sham-controlled, phase 3 trials. Lancet. 2023 Oct 21;402(10411):1434-1448. doi: 10.1016/S0140-6736(23)01520-9. PMID 37865470
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, randomized, double-masked, sham injection-controlled study was conducted in subjects with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) at 122 sites in 14 countries between 31 Aug 2018 and 20 Jun 2022.
Pre-assignment Details: This study consisted of a screening period (up to 30 days), a randomization visit on Day 1, and a treatment period (up to 24 months). Subjects were randomized in a 2:2:1:1 ratio on Day 1 to receive treatment with pegcetacoplan monthly, pegcetacoplan every other month (EOM), sham injection monthly or sham injection EOM, respectively. A total of 621 subjects were randomized in this study.
Groups:
- Pegcetacoplan Monthly: Subjects received intravitreal (IVT) injections of pegcetacoplan 15 milligram (mg)/0.1 milliliter (mL) once monthly for 24 months.
- Pegcetacoplan EOM: Subjects received IVT injections of pegcetacoplan 15 mg/0.1 mL EOM for 24 months.
- Sham Monthly: Subjects received sham injections once monthly for 24 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Sham EOM: Subjects received sham injections EOM for 24 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
Period: Overall Study
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Monthly | Sham EOM
Started | 206 | 208 | 102 | 105
Completed | 147 | 161 | 78 | 83
Not Completed | 59 | 47 | 24 | 22
Not completed — Adverse Event | 9 | 6 | 5 | 3
Not completed — Lost to Follow-up | 2 | 4 | 4 | 0
Not completed — Physician Decision | 1 | 0 | 2 | 0
Not completed — Consent withdrawal | 36 | 20 | 6 | 13
Not completed — Death | 7 | 6 | 4 | 3
Not completed — Due to Coronavirus Disease-2019 (COVID-19) impact | 4 | 10 | 3 | 3
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) analysis set consisted of all subjects assigned to treatment.
Groups:
- Pegcetacoplan Monthly: Subjects received IVT injections of pegcetacoplan 15 mg/0.1 mL once monthly for 24 months.
- Sham Pooled: Sham Monthly: Subjects received sham injections once monthly for 24 months.
  Sham EOM: Subjects received sham injections EOM for 24 months.
  The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Total: Total of all reporting groups
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled | Total
Number analyzed (Participants) | 206 | 208 | 207 | 621
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.8 (6.91) | 79.2 (7.06) | 78.5 (7.24) | 78.8 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 126 | 132 | 379
  Male | 85 | 82 | 75 | 242
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 192 | 192 | 200 | 584
  Not reported | 12 | 11 | 6 | 29
  Black or African American | 1 | 1 | 0 | 2
  Asian | 0 | 1 | 0 | 1
  Multiple | 0 | 1 | 0 | 1
  Unknown | 1 | 2 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 37 | 29 | 98
  Not Hispanic or Latino | 163 | 155 | 172 | 490
  Not Reported | 10 | 12 | 6 | 28
  Unknown | 1 | 4 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 146 | 126 | 128 | 400
  Argentina | 18 | 24 | 18 | 60
  France | 12 | 14 | 7 | 33
  Brazil | 9 | 13 | 10 | 32
  United Kingdom | 5 | 6 | 10 | 21
  Germany | 3 | 4 | 11 | 18
  Poland | 2 | 7 | 6 | 15
  Czechia | 2 | 7 | 5 | 14
  Australia | 3 | 1 | 4 | 8
  Canada | 2 | 1 | 4 | 7
  Israel | 0 | 4 | 2 | 6
  Italy | 2 | 1 | 0 | 3
  Spain | 1 | 0 | 2 | 3
  New Zealand | 1 | 0 | 0 | 1
GA Lesion Size (fundus autofluorescence [FAF]) in the Study Eye [Mean (Standard Deviation); unit: Millimeter square (mm^2)] | 8.3606 (4.16892) | 8.2076 (3.91213) | 8.2572 (4.21864) | 8.2749 (4.09557)

OUTCOME MEASURES:

1. Primary Outcome: Least Squares (LS) Mean Change From Baseline in Total Area of GA Lesions in the Study Eye at Month 12
Description: The GA lesion area was measured by a quantified central reading center based on FAF images. LS mean was calculated using a mixed effect model for repeated measure (MMRM) model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 12
Population: The modified ITT (mITT) analysis set consisted of all subjects assigned to treatment who received at least 1 injection of pegcetacoplan or sham and had baseline and at least 1 post-baseline value of GA lesion area in the study eye as assessed by FAF. Subjects with a baseline and at least 1 post-baseline value of the outcome at a scheduled visit by Month 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 200 | 199 | 193
mm^2 | 1.7344 (0.07924) | 1.7563 (0.07446) | 1.9640 (0.09592)
Statistical Analysis 1: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Model included treatment + baseline GA lesion area (<7.5 mm^2 or ≥7.5 mm^2) + analysis visit + presence of choroidal neovascularization (CNV) in the fellow eye (yes or no) + analysis visit × treatment + baseline GA lesion area × analysis visit; Test type: Superiority; p = 0.0615, MMRM model; LS Mean Difference = -0.2296, 95% CI 2-sided [-0.4703 to 0.0111]
Statistical Analysis 2: Comparison: Pegcetacoplan EOM vs Sham Pooled; Model included treatment + baseline GA lesion area (<7.5 mm^2 or ≥7.5 mm^2) + analysis visit + presence of CNV in the fellow eye (yes or no) + analysis visit × treatment + baseline GA lesion area × analysis visit; Test type: Superiority; p = 0.0854, MMRM model; LS Mean Difference = -0.2077, 95% CI 2-sided [-0.4444 to 0.0290]

2. Secondary Outcome: LS Mean Change From Baseline in the Total Area of GA Lesions in the Study Eye at Month 24
Description: The GA lesion area was measured by a quantified central reading center based on FAF images. LS mean was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: The mITT analysis set consisted of all subjects assigned to treatment who received at least 1 injection of pegcetacoplan or sham and had baseline and at least 1 post-baseline value of GA lesion area in the study eye as assessed by FAF. Subjects with a baseline and at least 1 post-baseline value of the outcome at a scheduled visit by Month 24 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 200 | 200 | 194
mm^2 | 3.2275 (0.12457) | 3.3395 (0.13034) | 3.9726 (0.16820)
Statistical Analysis 1: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Model included treatment + baseline GA lesion area (<7.5 mm^2 or ≥7.5 mm^2) + analysis visit + baseline presence of CNV in the fellow eye (yes or no) + analysis visit × treatment + baseline GA lesion area (<7.5 mm^2 or ≥7.5 mm^2) × analysis visit; Test type: Superiority; p = 0.0004, MMRM model; LS Mean Difference = -0.7451, 95% CI 2-sided [-1.1539 to -0.3362]
Statistical Analysis 2: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0030, MMRM model; LS Mean Difference = -0.6331, 95% CI 2-sided [-1.0508 to -0.2153]

3. Secondary Outcome: Mean Change in Total Area of GA Lesions in the Study Eye Through Month 24
Description: The mean change in GA lesion area through Month 24 was measured by assuming a piecewise linear trend in time with knots by FAF images at Months 6, 12, and 18 and was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: From Baseline (screening) through Month 24
Population: The mITT analysis set consisted of all subjects assigned to treatment who received at least 1 injection of pegcetacoplan or sham and had baseline and at least 1 post-baseline value of GA lesion area in the study eye as assessed by FAF.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 201 | 201 | 195
mm^2
  From Baseline to Month 6 | 0.9075 (0.04755) | 0.8829 (0.04660) | 0.9622 (0.04983)
  From Month 6 to Month 12 | 0.8409 (0.05128) | 0.8473 (0.05086) | 1.0132 (0.05998)
  From Month 12 to Month 18 | 0.9033 (0.04917) | 0.8803 (0.05105) | 1.0483 (0.05574)
  From Month 18 to Month 24 | 0.6262 (0.06809) | 0.6946 (0.05256) | 0.9794 (0.05469)
  From Baseline to Month 24 | 3.2780 (0.12525) | 3.3051 (0.12871) | 4.0031 (0.16880)
Statistical Analysis 1: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Baseline to Month 6: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — Baseline GA lesion area x Time (continuous) + Baseline GA lesion area x Time Spline at Month 6 (continuous) + Baseline GA lesion area x Time Spline at Month 12 (continuous) + Baseline GA lesion area x Time Spline at Month 18 (continuous). A heterogeneous autoregressive covariance matrix was used to model within-subject errors; p = 0.4282, MMRM model; Mean Difference = -0.0547, 95% CI 2-sided [-0.1899 to 0.0806]
Statistical Analysis 2: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.2457, MMRM model; Mean Difference = -0.0793, 95% CI 2-sided [-0.2131 to 0.0546]
Statistical Analysis 3: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Month 6 to Month 12: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0292, MMRM model; Mean Difference = -0.1722, 95% CI 2-sided [-0.3270 to -0.0174]
Statistical Analysis 4: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 3]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0352, MMRM model; Mean Difference = -0.1659, 95% CI 2-sided [-0.3202 to -0.0115]
Statistical Analysis 5: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Month 12 to Month 18: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0514, MMRM model; Mean Difference = -0.1450, 95% CI 2-sided [-0.2909 to 0.0009]
Statistical Analysis 6: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 5]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0265, MMRM model; Mean Difference = -0.1680, 95% CI 2-sided [-0.3164 to -0.0196]
Statistical Analysis 7: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Month 18 to Month 24: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM model; Mean Difference = -0.3532, 95% CI 2-sided [-0.5245 to -0.1819]
Statistical Analysis 8: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 7]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0002, MMRM model; Mean Difference = -0.2848, 95% CI 2-sided [-0.4336 to -0.1361]
Statistical Analysis 9: Comparison: Pegcetacoplan Monthly vs Sham Pooled; Estimates for Baseline to Month 24: Model included Treatment + Baseline GA lesion area (< 7.5 mm^2 or >= 7.5 mm^2) + Time (continuous) + Time Spline at Month 6 (continuous) + Time Spline at Month 12 (continuous) + Time Spline at Month 18 (continuous) + Presence of CNV in the fellow eye (Yes or No) + Time (continuous) x Treatment + Time Spline at Month 6 (continuous) x Treatment + Time Spline at Month 12 (continuous) x Treatment + Time Spline at Month 18 (continuous) x Treatment +; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0006, MMRM model; Mean Difference = -0.7251, 95% CI 2-sided [-1.1373 to -0.3129]
Statistical Analysis 10: Comparison: Pegcetacoplan EOM vs Sham Pooled; [analysis description as in outcome 3, analysis 9]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0010, MMRM model; Mean Difference = -0.6980, 95% CI 2-sided [-1.1142 to -0.2817]

4. Secondary Outcome: LS Mean Change From Baseline in Monocular Maximum Reading Speed of the Study Eye at Month 24
Description: The maximum reading speed of the study eye was calculated per Minnesota Low-Vision Reading Test (MNREAD) or Radner Reading Charts user manuals, with no adjustment for reading inaccuracy. An additional step to cap resulting reading speed values at a maximum of 300 words per minute (wpm) was implemented. Maximum reading speed was calculated as the mean of the 3 highest non-zero reading speeds (or 2, or 1 value, as available), except when all wpm were calculated as 0 then the maximum reading speed was calculated as 0. LS mean was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: wpm
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 179 | 163 | 164
wpm | -22.897 (4.1171) | -25.532 (2.7676) | -22.355 (2.9341)

5. Secondary Outcome: LS Mean Change From Baseline in Mean Functional Reading Independence (FRI) Index Score at Month 24
Description: The FRI was an interviewer-administered questionnaire with 7 items on functional reading activities most relevant to GA AMD subjects. It had 1 total index score. For each FRI Index reading activity performed in the past 7 days, subjects were asked about the extent to which they required assistance beyond eyeglasses/contact lenses, including the use of low-vision aids, adjustments in the activity, or help from another subject. Mean FRI Index scores ranged from 1 (unable to do independently) to 4 (totally independent), with higher scores indicating higher functional reading independence. A negative change from baseline indicated a decrease in the FRI; disease worsening. LS mean was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 186 | 183 | 178
scores on a scale | -0.408 (0.0570) | -0.371 (0.0562) | -0.360 (0.0601)

6. Secondary Outcome: LS Mean Change From Baseline in Normal-Luminance Best-Corrected Visual Acuity (NL-BCVA) Score of the Study Eye at Month 24
Description: The NL-BCVA was assessed by early treatment diabetic retinopathy study (ETDRS) chart prior to dilating the eyes at a starting distance of 4 meters and ranged from 0 (least score) to 100 (best score). If the 4-meter score was >19 letters read correctly, the visual acuity score was the sum of total letters correctly read at 4 meters plus the addition of 30. If the 4-meter score was ≤19 letters read correctly, the visual acuity score was the sum of total letters read correctly at 4 meters and total letters read correctly at the 1-meter distance. If no letters were read correctly at either the 4-meter distance or the 1-meter distance, the visual acuity score was 0. A positive change in the value indicated improvement in visual acuity. LS mean was calculated using a MMRM model. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ETDRS letter score
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 201 | 201 | 195
ETDRS letter score | -8.126 (1.0182) | -8.947 (1.0322) | -6.217 (1.0167)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were reported from first study drug administration (Day 1) up to the last visit or early termination visit, 30 days after the last study drug administration for the monthly treatment groups and 60 days after the last study drug administration for the EOM treatment groups, a maximum of 24 months
Description: The Safety analysis set consisted of all randomized subjects who received at least 1 injection of pegcetacoplan or sham. Ocular TEAEs are presented separately for the study and fellow eyes, and non-ocular (systemic) TEAEs are also presented.
Groups:
- Pegcetacoplan Monthly: Ocular Study Eye: Ocular TEAEs were summarized for the study eye for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL once monthly for 24 months.
- Pegcetacoplan EOM: Ocular Study Eye: Ocular TEAEs were summarized for the study eye for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL EOM for 24 months.
- Sham Pooled: Ocular Study Eye: Ocular TEAEs were summarized for the study eye for all subjects who were randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 24 months.
  Sham EOM: Subjects received sham injections EOM for 24 months.
  The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Pegcetacoplan Monthly: Ocular Fellow Eye: Ocular TEAEs were summarized for the fellow eye for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL once monthly for 24 months.
- Pegcetacoplan EOM: Ocular Fellow Eye: Ocular TEAEs were summarized for the fellow eye for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL EOM for 24 months.
- Sham Pooled: Ocular Fellow Eye: Ocular TEAEs were summarized for the fellow eye for all subjects who were randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 24 months.
  Sham EOM: Subjects received sham injections EOM for 24 months.
  The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Pegcetacoplan Monthly: Non-ocular: Non-ocular (systemic) TEAEs were summarized for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL once monthly for 24 months.
- Pegcetacoplan EOM: Non-ocular: Non-ocular (systemic) TEAEs were summarized for all subjects who received IVT injections of pegcetacoplan 15 mg/0.1 mL EOM for 24 months.
- Sham Pooled: Non-ocular: Non-ocular (systemic) TEAEs were summarized for all subjects who were randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 24 months.
  Sham EOM: Subjects received sham injections EOM for 24 months.
  The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
Arm/Group | Pegcetacoplan Monthly: Ocular Study Eye | Pegcetacoplan EOM: Ocular Study Eye | Sham Pooled: Ocular Study Eye | Pegcetacoplan Monthly: Ocular Fellow Eye | Pegcetacoplan EOM: Ocular Fellow Eye | Sham Pooled: Ocular Fellow Eye | Pegcetacoplan Monthly: Non-ocular | Pegcetacoplan EOM: Non-ocular | Sham Pooled: Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/208 | 0/206 | 0/206 | 0/208 | 0/206 | 8/206 | 6/208 | 8/206
Serious Adverse Events (participants affected / at risk) | 4/206 | 2/208 | 2/206 | 1/206 | 1/208 | 0/206 | 61/206 | 47/208 | 53/206
Other Adverse Events (participants affected / at risk) | 113/206 | 82/208 | 61/206 | 35/206 | 34/208 | 29/206 | 90/206 | 70/208 | 101/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegcetacoplan Monthly: Ocular Study Eye (N=206) | Pegcetacoplan EOM: Ocular Study Eye (N=208) | Sham Pooled: Ocular Study Eye (N=206) | Pegcetacoplan Monthly: Ocular Fellow Eye (N=206) | Pegcetacoplan EOM: Ocular Fellow Eye (N=208) | Sham Pooled: Ocular Fellow Eye (N=206) | Pegcetacoplan Monthly: Non-ocular (N=206) | Pegcetacoplan EOM: Non-ocular (N=208) | Sham Pooled: Non-ocular (N=206)
Uveitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitritis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathogen resistance (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Superficial spreading melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegcetacoplan Monthly: Ocular Study Eye (N=206) | Pegcetacoplan EOM: Ocular Study Eye (N=208) | Sham Pooled: Ocular Study Eye (N=206) | Pegcetacoplan Monthly: Ocular Fellow Eye (N=206) | Pegcetacoplan EOM: Ocular Fellow Eye (N=208) | Sham Pooled: Ocular Fellow Eye (N=206) | Pegcetacoplan Monthly: Non-ocular (N=206) | Pegcetacoplan EOM: Non-ocular (N=208) | Sham Pooled: Non-ocular (N=206)
Vitreous floaters (Eye disorders) | 24 (29) | 10 (12) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 21 (22) | 10 (10) | 5 (6) | 7 (8) | 11 (11) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 12 (16) | 15 (21) | 5 (6) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 9 (9) | 15 (15) | 8 (9) | 2 (3) | 4 (5) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 16 (16) | 6 (8) | 10 (11) | 10 (11) | 6 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 8 (8) | 14 (14) | 6 (6) | 8 (8) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 13 (18) | 8 (9) | 13 (15) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 8 (8) | 12 (12)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (12) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 17 (30) | 13 (15) | 21 (36)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 7 (7) | 11 (11)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (16) | 15 (20) | 21 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 4 (5) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (16) | 6 (8) | 14 (16)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 17 (18) | 16 (16) | 15 (15)
Eye irritation (Eye disorders) | 10 (13) | 4 (5) | 11 (12) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT03525600/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03525600/SAP_001.pdf